CLINICAL TRIAL: NCT05030870
Title: Capnographic Monitoring Decrease the Incidence of Hypoxia of the Elderly Patients Undergoing Gastrointestinal Endoscopy Procedure: a Randomized Multicenter Clinical Trial
Brief Title: Capnographic Monitoring in Gastrointestinal Endoscopy for Elderly Patients
Acronym: CapnoGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Henan Provincial People's Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RenjiH-20201201
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypoxia; Gastric Cancer; Gastric Polyp; Colon Polyp; Colon Cancer; Esophageal Cancer
Keywords: Capnographic Monitoring; Hypoxia; Gastrointestinal endoscopy; Elderly patients; Propofol
MeSH Terms: conditions — Hypoxia; Stomach Neoplasms; Polyposis, Gastric; Colonic Polyps; Colonic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capnographic monitoring group (Experimental): In this group, in addition to the standard monitoring including observation, pulse oxygen saturation, non-invasive blood pressure, electrocardiogram in selected patients, the capnographic is also monitored. The capnographic data of the patients are available for additional noninvasive assessment of ventilation.
  Interventions: Device: Capnography monitoring; Device: Standard monitoring
- Standard monitoring group (Active Comparator): In this group, standard monitoring including observation, pulse oxygen saturation, non-invasive blood pressure, electrocardiogram in selected patients. Capnographic data are not visible by closing the CO2 sampling line till the endoscopy end.
  Interventions: Device: Standard monitoring

INTERVENTIONS:
Device: Capnography monitoring — Standard monitoring and capnographic monitoring.
  Arms: Capnographic monitoring group
Device: Standard monitoring — Standard monitoring but no capnographic monitoring

SUMMARY:
Hypoxia is the most common adverse event in gastrointestinal endoscopes sedated with propofol and sufentanil, especially in elderly people. The aim of this randomized study was to determine whether intervention based on additional capnographic monitoring reduces the incidence of hypoxia in gastrointestinal endoscopes procedures for elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 ≤ Age <80
* patients undergoing gastrointestinal endoscopes
* patients signed informed consent form
* ASA classification I-II

Exclusion Criteria:

* Coagulation disorders or a tendency of nose bleeding
* An episode/exacerbation of congestive heart failure (CHF) that requires a change in medication, diet or hospitalization from any cause in the last 6 months
* Severe aortic stenosis or mitral stenosis
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months
* Acute myocardial infarction in the last 6 months
* Acute arrhythmia (including any tachycardia - or bradycardia) with the fluid of hemodynamics instability
* Diagnosed chronic obstructive pulmonary disease or current other acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy)
* Pre-existing bradycardia (heart rate < 50 / min), or hypoxia (SaO2< 90 % )
* Need supplemental oxygen because of pre-existing diseases
* Emergency procedure or surgery
* Multiple trauma
* Upper respiratory tract infection
* Allergy to propofol or tape and adhesives

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (75% ≤ SpO2 < 90% for <60 s)

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (90% ≤ SpO2 < 95%)
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (SpO2 < 75% or 75% ≤ SpO2 < 90% for >/=60 s)
The incidence of capnography curve decreased by half or more than the baseline and even disappeared without hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  capnography curve decreased by half or more than the baseline and even disappeared, SpO2 >90%
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Principal Investigator — Department of Anesthesiology Renji Hospital
Locations (3):
- China (3):
  - Henan Provincial People's Hospital, Zhenzhou, Henan
  - Qilu Hospital of Shandong University, Qingdao, Shandong
  - Renji Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Lian Q, Chen S, Cheng X, Zhang J, Yu W, Zhou R, Su D. Capnographic monitoring reduces hypoxia incidence in older patients undergoing gastrointestinal endoscopy under propofol sedation: study protocol for a multicenter randomized controlled trial. Trials. 2023 Mar 15;24(1):192. doi: 10.1186/s13063-023-07208-0. PMID 36918924